CLINICAL TRIAL: NCT00805064
Title: Intravitreal Combination Therapy Using Triamcinolone and Bevacizumab Improves Vision in Patients With Retinal Vein Occlusion
Brief Title: Combined Triple Procedure in Retinal Vein Occlusion (RVO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Michael Koss, PI, Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-KTRVO-2008
Record Dates: First submitted 2008-12-04; First posted 2008-12-09 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Triamcinolone; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ischemic CRVO (Active Comparator): treatment was applied to this entity
  Interventions: Drug: triamcinolone and bevacizumab
- non ischemic CRVO (Active Comparator): treatment was applied to this entity
  Interventions: Drug: triamcinolone and bevacizumab
- BRVO (Active Comparator): treatment was applied to this entity
  Interventions: Drug: triamcinolone and bevacizumab

INTERVENTIONS:
Drug: triamcinolone and bevacizumab

SUMMARY:
The aim of this pilot study was to investigate the effects of an intravitreal combination therapy using triamcinolone and bevacizumab in patients with retinal vein occlusion (RVO).

DETAILED DESCRIPTION:
This prospective study of a case series was conducted in 47 patients (n = 47 eyes; f/m: 21/26; mean age: 66.6 years) with ischemic central RVO (CRVO) (n = 15), non-ischemic CRVO (n = 7), or branch RVO (BRVO) (n = 25). A core pars plana vitrectomy with aspiration of 1.5 ml vitreous and infusion of balanced salt solution (BSS; 1 ml), 8 mg (0.4 ml) triamcinolone, and 1.25 mg (0.1 ml) bevacizumab was performed with a single sutureless sclerotomy and a 23 gauge probe tip. At baseline and follow-up, the best corrected visual acuity (BCVA; 6 m Snellen), and intraocular pressure (IOP; Goldmann tonometry), and central macular thickness (optical coherence tomography) were determined. In addition, the need for further treatment and adverse events were monitored.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic central RVO (CRVO)
* Non-ischemic CRVO
* Branch RVO (BRVO)

Exclusion Criteria:

* Visual deterioration due to acute or chronic inflammation
* Post trauma
* Macular edema of other origin
* Intravitreal drug treatment within last 4 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
BCVA | day of exam

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koss, MD, Principal Investigator — Department of VitreoRetinal Surgery ZAU JWGU